CLINICAL TRIAL: NCT05288751
Title: Contingency Management as a Treatment for Opioid Use Disorder and Stimulant Use Disorder in a Primary Care Setting
Brief Title: Contingency Management for Opioid and Stimulant Use Disorders in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FMCH-2022-30581
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder; Stimulant Use Disorder
Keywords: opioid use disorder; stimulant use disorder; contingency management; primary care; addiction medicine; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (TAU) (No Intervention): These patients will not be assigned to the CM programs, but will be invited to complete study measures at the same time points: baseline, 3-months, 6-months, and 12-months.
- Attendance-only CM (Experimental): Patients in this arm complete an appointments with his or her primary care provider (PCP) or member of the PCP's microteam . These appointments must be initiated by the PCP/microteam in accordance with the patient's treatment plan for regular follow-up appointments.
  Interventions: Behavioral: Contingency Management
- Attendance + abstinence CM (Experimental): Patients who test stimulant-positive during the initial urine drug screen (UDS) at their intake visit will be invited to additionally enroll in the abstinence CM schedule. All of the attendance-only CM rules described previously will apply to patients in the attendance + abstinence program.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management (CM) is a behavioral intervention that involves incentivizing participants for target behaviors in a clinical setting.
  Arms: Attendance + abstinence CM; Attendance-only CM

SUMMARY:
Contingency management (CM) is a behavioral intervention that involves incentivizing participants for target behaviors in a clinical setting. When applied to the treatment of substance use disorders, it has demonstrated efficacy in reducing the number of urine toxicology screens positive for illicit substances and increased engagement in treatment programs. However, there is a need to translate CM treatment to primary care settings. This study will implement and assess a CM program for patients with opioid use disorder, with or without comorbid stimulant use disorder, initiating outpatient addiction medicine services at a family medicine residency clinic. Eligible patients will earn monetary incentives for attending addiction medicine appointments and abstaining from substances during outpatient treatment. Data gathered from this pilot program will be used to improve patient outcomes, treatment, and retention for persons receiving medications for opioid use disorder (MOUDs) in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of Opioid Use Disorder and/or Stimulant Use Disorder
* Recently initiated medications for opioid use disorder (MOUDs) at Broadway Family Medicine (BFM), within 2 weeks of recruitment
* Have an active prescription for buprenorphine-naloxone (Suboxone)

Exclusion Criteria:

* Prescription for an amphetamine would exclude patients from the abstinence-based CM, but they could participate in the attendance-only CM.
* Dementia, development disabilities, or cognitive functioning that is too low to participate in study measures, as determined by chart review and consultation with overseeing physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Preliminary efficacy of CM on clinical outcomes: Visit Frequency | 30 days post-intervention
  Number of completed clinical visits per patient during the CM program.
Preliminary efficacy of CM on clinical outcomes: Urine toxicology | 30 days post-intervention
  Percentage of UDS results that are negative for stimulants during the CM intervention period.
Feasibility of CM for OUD in primary care: Recruitment | 30 days post-intervention
  percentage of patients invited to participate enroll in the treatment intervention.
Feasibility of CM for OUD in primary care: Retention | 30 days post-intervention
  Of those patients who enroll in the intervention study, the percent that complete the CM intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levy, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States